CLINICAL TRIAL: NCT00077831
Title: Neurobehavioral Correlates of Craniosynostosis
Brief Title: Child and Infant Learning Project
Acronym: CILP
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Matt Speltz, Principal Investigator, Seattle Children's Hospital
Other Study IDs: NIDCR-13813; R01DE013813 (NIH)
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Craniosynostosis
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: neurobehavioral development — observational study of infant and child development

SUMMARY:
To learn more about the cognitive and motor development of infants and young children born with a craniofacial defect called craniosynostosis.

DETAILED DESCRIPTION:
In the first phase of this multi-site, 10-year longitudinal study, infants with one of four types of single-suture craniosynostosis were recruited: sagittal, metopic, right unilateral coronal, and left unilateral coronal. A case-matched "control" group of healthy, normal infants was also followed. This study, which is now in its second phase, is following this same cohort of children at the age of 7 years.

ELIGIBILITY:
Enrollment criteria at Phase 1:

* Confirmed diagnosis of single-suture, nonsyndromic craniosynostosis (sagittal, metopic, unilateral coronal, or lambdoid)
* Corrective (cranioplastic) surgery not yet performed
* Child born at 34 weeks gestation or later
* Absence of neurological conditions/significant health problems
* 33 months or younger at time of enrollment (male or female).

Enrollment criteria at Phase 2:

All participants enrolled in phase 1 are invited to participate in phase 2.

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with single-suture craniosynostosis between the ages of 2 months and 3 years were recruited and followed during phase 1. This same chort of children are now being followed at the age of 7 (phase 2). See eligibility criteria section for more information.
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2001-09; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopment as assessed by the Bayley Scales of Infant Development II | 1st assessment - post diagnosis, pre surgery. 2nd assessment - Target age 18 months. 3rd assessment - Target age 36 months.

SECONDARY OUTCOMES:
Neurodevelopment as assessed by the Wechsler Intelligence Scale for Children Version IV | Target age 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L. Speltz, Principal Investigator — Seattle Children's Hospital
Locations (4):
- United States (4):
  - Children's Health Care of Atlanta, Atlanta, Georgia
  - Northwestern University, Cleft Lip and Palate Institute, Westchester, Illinois
  - St. Louis Children's Hospital / Washington University, St Louis, Missouri
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Background] Speltz ML, Kapp-Simon KA, Cunningham M, Marsh J, Dawson G. Single-suture craniosynostosis: a review of neurobehavioral research and theory. J Pediatr Psychol. 2004 Dec;29(8):651-68. doi: 10.1093/jpepsy/jsh068. PMID 15491988
- [Background] McCarthy JG, Warren SM, Bernstein J, Burnett W, Cunningham ML, Edmond JC, Figueroa AA, Kapp-Simon KA, Labow BI, Peterson-Falzone SJ, Proctor MR, Rubin MS, Sze RW, Yemen TA; Craniosynostosis Working Group. Parameters of care for craniosynostosis. Cleft Palate Craniofac J. 2012 Jan;49 Suppl:1S-24S. doi: 10.1597/11-138. Epub 2011 Aug 17. PMID 21848431
- [Result] Starr JR, Kapp-Simon KA, Cloonan YK, Collett BR, Cradock MM, Buono L, Cunningham ML, Speltz ML. Presurgical and postsurgical assessment of the neurodevelopment of infants with single-suture craniosynostosis: comparison with controls. J Neurosurg. 2007 Aug;107(2 Suppl):103-10. doi: 10.3171/PED-07/08/103. PMID 18459881
- [Result] Lin HJ, Ruiz-Correa S, Shapiro LG, Speltz ML, Cunningham ML, Sze RW. Predicting neuropsychological development from skull imaging. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:3450-5. doi: 10.1109/IEMBS.2006.260321. PMID 17945777
- [Result] Ruiz-Correa S, Starr JR, Lin HJ, Kapp-Simon KA, Cunningham ML, Speltz ML. Severity of skull malformation is unrelated to presurgery neurobehavioral status of infants with sagittal synostosis. Cleft Palate Craniofac J. 2007 Sep;44(5):548-54. doi: 10.1597/06-190.1. PMID 17760493
- [Result] Toth K, Collett B, Kapp-Simon KA, Cloonan YK, Gaither R, Cradock MM, Buono L, Cunningham ML, Dawson G, Starr J, Speltz ML. Memory and response inhibition in young children with single-suture craniosynostosis. Child Neuropsychol. 2008 Jul;14(4):339-52. doi: 10.1080/09297040701594888. Epub 2007 Sep 26. PMID 17899471
- [Result] Kapp-Simon KA, Speltz ML, Cunningham ML, Patel PK, Tomita T. Neurodevelopment of children with single suture craniosynostosis: a review. Childs Nerv Syst. 2007 Mar;23(3):269-81. doi: 10.1007/s00381-006-0251-z. Epub 2006 Dec 21. PMID 17186250
- [Result] Kapp-Simon KA, Leroux B, Cunningham M, Speltz ML. Multisite study of infants with single-suture craniosynostosis: preliminary report of presurgery development. Cleft Palate Craniofac J. 2005 Jul;42(4):377-84. doi: 10.1597/04-044.1. PMID 16001919
- [Result] Ruiz-Correa S, Sze RW, Starr JR, Lin HT, Speltz ML, Cunningham ML, Hing AV. New scaphocephaly severity indices of sagittal craniosynostosis: a comparative study with cranial index quantifications. Cleft Palate Craniofac J. 2006 Mar;43(2):211-21. doi: 10.1597/04-208.1. PMID 16526927
- [Result] Cunningham ML, Horst JA, Rieder MJ, Hing AV, Stanaway IB, Park SS, Samudrala R, Speltz ML. IGF1R variants associated with isolated single suture craniosynostosis. Am J Med Genet A. 2011 Jan;155A(1):91-7. doi: 10.1002/ajmg.a.33781. PMID 21204214
- [Result] Kapp-Simon KA, Collett BR, Barr-Schinzel MA, Cradock MM, Buono LA, Pietila KE, Speltz ML. Behavioral adjustment of toddler and preschool-aged children with single-suture craniosynostosis. Plast Reconstr Surg. 2012 Sep;130(3):635-647. doi: 10.1097/PRS.0b013e31825dc18b. PMID 22929249
- [Result] Mefford HC, Shafer N, Antonacci F, Tsai JM, Park SS, Hing AV, Rieder MJ, Smyth MD, Speltz ML, Eichler EE, Cunningham ML. Copy number variation analysis in single-suture craniosynostosis: multiple rare variants including RUNX2 duplication in two cousins with metopic craniosynostosis. Am J Med Genet A. 2010 Sep;152A(9):2203-10. doi: 10.1002/ajmg.a.33557. PMID 20683987
- [Result] Naumann HL, Haberkern CM, Pietila KE, Birgfeld CB, Starr JR, Kapp-Simon KA, Hopper RA, Speltz ML. Duration of exposure to cranial vault surgery: associations with neurodevelopment among children with single-suture craniosynostosis. Paediatr Anaesth. 2012 Nov;22(11):1053-61. doi: 10.1111/j.1460-9592.2012.03843.x. PMID 22502768
- [Result] Rosenberg JM, Kapp-Simon KA, Starr JR, Cradock MM, Speltz ML. Mothers' and fathers' reports of stress in families of infants with and without single-suture craniosynostosis. Cleft Palate Craniofac J. 2011 Sep;48(5):509-18. doi: 10.1597/09-210. Epub 2010 Aug 19. PMID 20815729
- [Result] Ruiz-Correa S, Starr JR, Lin HJ, Kapp-Simon KA, Sze RW, Ellenbogen RG, Speltz ML, Cunningham ML. New severity indices for quantifying single-suture metopic craniosynostosis. Neurosurgery. 2008 Aug;63(2):318-24; discussion 324-5. doi: 10.1227/01.NEU.0000316417.06500.DA. PMID 18797362
- [Result] Seto ML, Hing AV, Chang J, Hu M, Kapp-Simon KA, Patel PK, Burton BK, Kane AA, Smyth MD, Hopper R, Ellenbogen RG, Stevenson K, Speltz ML, Cunningham ML. Isolated sagittal and coronal craniosynostosis associated with TWIST box mutations. Am J Med Genet A. 2007 Apr 1;143A(7):678-86. doi: 10.1002/ajmg.a.31630. PMID 17343269
- [Result] Speltz ML, Kapp-Simon K, Collett B, Keich Y, Gaither R, Cradock MM, Buono L, Cunningham ML. Neurodevelopment of infants with single-suture craniosynostosis: presurgery comparisons with case-matched controls. Plast Reconstr Surg. 2007 May;119(6):1874-1881. doi: 10.1097/01.prs.0000259184.88265.3f. PMID 17440368
- [Result] Starr JR, Collett BR, Gaither R, Kapp-Simon KA, Cradock MM, Cunningham ML, Speltz ML. Multicenter study of neurodevelopment in 3-year-old children with and without single-suture craniosynostosis. Arch Pediatr Adolesc Med. 2012 Jun 1;166(6):536-42. doi: 10.1001/archpediatrics.2011.1800. PMID 22312170
- [Result] Starr JR, Lin HJ, Ruiz-Correa S, Cunningham ML, Ellenbogen RG, Collett BR, Kapp-Simon KA, Speltz ML. Little evidence of association between severity of trigonocephaly and cognitive development in infants with single-suture metopic synostosis. Neurosurgery. 2010 Aug;67(2):408-15; discussion 415-6. doi: 10.1227/01.NEU.0000371992.72539.8B. PMID 20644427
- [Result] Collett BR, Gray KE, Kapp-Simon KA, Birgfeld C, Cunningham M, Rudo-Stern J, Ung D, Buono L, Speltz ML. Laypersons' ratings of appearance in children with and without single-suture craniosynostosis. J Craniofac Surg. 2013 Jul;24(4):1331-5. doi: 10.1097/SCS.0b013e3182997885. PMID 23851801
- [Result] Gray KE, Cradock MM, Kapp-Simon KA, Collett BR, Pullmann LD, Speltz ML. Longitudinal analysis of parenting stress in mothers and fathers of infants with and without single-suture craniosynostosis. Cleft Palate Craniofac J. 2015 Jan;52(1):3-11. doi: 10.1597/13-239. PMID 24841516